CLINICAL TRIAL: NCT00383513
Title: An Open-Label Re-treatment Trial for Patients Previously Randomized Into the SL0003 and SL0004, Randomized, Double-blind, Placebo-controlled, Multi-center Studies of Epratuzumab in Patients With Systemic Lupus Erythematosus
Brief Title: Study of Epratuzumab in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL0006; EudraCT #: 2006-004496-36
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Antibody; B-Cell Immunotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epratuzumab (Experimental)
  Interventions: Biological: Epratuzumab

INTERVENTIONS:
Biological: Epratuzumab — 360 mg/m^2 four consecutive 12-week maintenance cycles beginning with 2 consecutive weekly administrations each lasting ≤ 1 hour

SUMMARY:
Epratuzumab is an investigational antibody designed to help treat Systemic Lupus Erythematosus (SLE). The purpose of the study is to obtain additional long-term information regarding the safety and efficacy of continued maintenance-cycle administrations of Epratuzumab.

DETAILED DESCRIPTION:
Due to the logistical considerations, UCB has decided to consolidate the Phase II and Phase III open-label extension trials. Subjects completing this study will be offered the option of continuing to receive epratuzumab through participation in Phase III open-label extension study SL0012 (NCT01408576).

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in SL0003 or SL0004 and benefitted from participation in those studies

Exclusion Criteria:

* Development of toxicity to epratuzumab
* Significant protocol deviations during the SL0003 or SL0004 studies
* Evidence of significant infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting at least 1 serious adverse event (SAE) from entry Visit 1 through end of treatment (approximately 6 years) | From Entry Visit 1 through end of treatment (approximately 6 years)
Number of subjects prematurely discontinuing due to a treatment emergent adverse event (TEAE) from entry Visit 1 through end of treatment (approximately 6 years) | From Entry Visit 1 through end of treatment (approximately 6 years)

SECONDARY OUTCOMES:
Time to treatment failure from First Visit through end of treatment (approximately 6 years) | From the first infusion of the first treatment cycle and continuing through end of treatment (approximately 6 years)
  Treatment failure is defined as initiation of a protocol specified prohibited medication.
Epratuzumab plasma concentration levels at Week 0 | Week 0
Epratuzumab plasma concentration levels at Week 48 | Week 48
Epratuzumab plasma concentration levels at Week 96 | Week 96
Epratuzumab plasma concentration levels at Week 144 | Week 144
Epratuzumab plasma concentration levels at Week 192 | Week 192
Epratuzumab plasma concentration levels at Week 240 | Week 240
Subject Epratuzumab plasma concentration levels at Week 288 | Week 288
Number of subjects with anti-epratuzumab antibody in plasma at Week 0 | Week 0
Number of subjects with anti-epratuzumab antibody in plasma at Week 48 | Week 48
Number of subjects with anti-epratuzumab antibody in plasma at Week 96 | Week 96
Number of subjects with anti-epratuzumab antibody in plasma at Week 144 | Week 144
Number of subjects with anti-epratuzumab antibody in plasma at Week 192 | Week 192
Number of subjects with anti-epratuzumab antibody in plasma at Week 240 | Week 240
Number of subjects with anti-epratuzumab antibody in plasma at Week 288 | Week 288
Change From Baseline in Short Form 36-items Health Survey (SF-36) Physical Component Summary (PCS) Score | Baseline, Last Visit
Change from Baseline in Short Form 36-items Health Survey (SF-36) Mental Composite Summary (MCS) Score | Baseline, Last Visit
Change from Baseline in Patient's Global Assessment of Disease Activity (PtGADA) | Baseline, Last Visit
  Five point scale where 1 = very poor and 5 = very good.
Change from Baseline in Physician's Global Assessment of Disease Activity (PGADA) | Baseline, Last Visit
  Five point scale where 1 = very poor and 5 = very good.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (10):
- United States (10):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Upland, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Baltimore, Maryland
  - Durham, North Carolina
  - Tulsa, Oklahoma